CLINICAL TRIAL: NCT07217808
Title: Precision-Medicine Diagnostic Support in Hospitalized Veterans With Acute Kidney Injury
Acronym: PRECISE-AKI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Tennessee Valley Health Care System (U.S. Federal Agency); Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: HSR3-017-24W
Record Dates: First submitted 2025-10-06; First posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Acute Kidney Injury (AKI)
Keywords: Acute Kidney Injury; Decision Support Systems, Clinical; Artificial Intelligence
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: Pre-/Post- design
Who Masked: Outcomes Assessor
Masking Description: It is not possible to blind clinicians. Study data will be extracted by staff blinded to assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Usual Care) (No Intervention): The Control arm will consist of usual care with no additional clinical decision support tool guidance
- PRECISION AKI Clinical Decision Support (Experimental): The Intervention arm will consist of Clinical Decision Diagnostic Support (CDS) provided by the PRECISE-AKI tool
  Interventions: Other: PRECISE-AKI Clinical Decision Support Tool

INTERVENTIONS:
Other: PRECISE-AKI Clinical Decision Support Tool — The Intervention arm will consist of Clinical Decision Diagnostic Support (CDS) provided by the PRECISE-AKI tool
  Arms: PRECISION AKI Clinical Decision Support

SUMMARY:
Acute kidney injury (AKI) affects up to 20% of hospitalized Veterans and is strongly associated with morbidity and death. AKI is a diverse condition and timely and accurate diagnosis of the type of AKI is critical to begin appropriate therapies, especially those causes that require specific treatments beyond general supportive care. Yet, there are still significant gaps in the initial evaluation of AKI among hospitalized patients. Clinical decision support systems (CDSS) have shown promise to address these barriers, but most consist of simple alerting schemes and general care recommendations provided at a single point in time. The goal of this proposal is to develop and test the feasibility and usability of a rule-based and Artificial Intelligence-assisted precision CDSS tool (PRECISE-AKI) that can provide cognitive support to improve timely initial diagnostic evaluation of AKI.

DETAILED DESCRIPTION:
Acute kidney injury (AKI), defined as a sudden loss of kidney function, affects up to 20% of hospitalized Veterans and is strongly associated with chronic kidney disease, poor quality of life, and death. Clinical practice guidelines recommend timely identification of the cause of AKI, but gaps remain in conducting the initial and subsequent diagnostic evaluation. Some causes of AKI also require specific treatments beyond supportive care, can be challenging to diagnose, and can require even more detailed evaluation including kidney biopsies. This clinical trial will evaluate the usability and feasibility of an Artificial Intelligence (AI)-assisted automated and comprehensive precision CDSS tool (PRECISE-AKI) to provide iterative cognitive support of general and nephrology-based providers in the diagnostic evaluation of hospitalized patients experiencing AKI within the Tennessee Valley Health Systems (TVHS). The investigators hypothesize that PRECISE-AKI will be acceptable, appropriate, and feasible to a variety of users and improve the diagnostic evaluation of hospitalized patients AKI.

ELIGIBILITY:
Inclusion Criteria:

* Eligible providers will be those that have at least 4 weeks of inpatient ward team or consultation team activity during a 12-month period.
* Case inclusion criteria will consist of hospitalizations that meet criteria for Kidney Disease Improving Global Outcomes Stage 2 injury or persistent Stage 1 injury seen by eligible providers.

Exclusion Criteria:

* Ineligible providers will be those that have < 4 weeks of inpatient ward team of consultative team activity during a 12 month period.
* Hospitalizations with non-persistent (<48 hours) stage 1 injury or less.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2028-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Rates of Appropriate Diagnostic Testing | Up to 30 days
  Based on the presenting context, the investigators will compare rates of appropriate diagnostic testing between intervention and control patients among those meeting the AKI case definition

OTHER OUTCOMES:
Exploratory Clinical Outcome: Peak Kidney Disease Improving Global Outcomes (KDIGO) AKI Stage during hospitalization. | During Index Hospitalization through 30 days
  For this exploratory clinical outcome, we will compare differences in the peak KDIGO AKI Stage (creatinine-based criteria) during hospitalization after meeting the case definition of AKI between intervention and control cases.
Exploratory Clinical Outcome: Discharge serum creatinine | Last serum creatinine during index hospitalization through 30 days
  The investigators will compare differences in the hospital discharge serum creatinine after meeting the case definition of AKI between intervention and control cases.
Exploratory Clinical Outcome: Major Adverse Kidney Events (MAKE) 90 | 90 days
  For this exploratory clinical outcome, the investigators will compare the rates of the major adverse kidney events experienced by eligible AKI cases in the intervention compared with the control arm. Major Adverse Kidney Events will be defined as kidney replacement therapy, death, or an increase in baseline serum creatinine of 150% of baseline using the last serum creatinine available up to 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Edward D Siew, MD MSc, Principal Investigator — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN; Michael E Matheny, MD MS MPH, Principal Investigator — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN
Locations (1):
- Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No